CLINICAL TRIAL: NCT00548587
Title: A Randomised, Double-Blind, Placebo-Controlled Study of the Safety and Tolerability of E5555, and Its Effects on Clinical Events and Biomarkers in Patients With Non-ST-Segment Elevation Acute Coronary Syndrome
Brief Title: Safety and Tolerability of E5555 and Its Effects on Markers of Intravascular Inflammation in Subjects With Acute Coronary Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E5555-G000-202; 2006-000296-15 (EudraCT Number)
Record Dates: First submitted 2007-10-22; First posted 2007-10-24 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2015-11

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — E 5555

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): Participants will receive one 50 mg E5555 tablet and two 100 mg placebo tablets, once daily for 12 weeks.
  Interventions: Drug: E5555; Drug: Placebo
- 2 (Active Comparator): Participants will receive one 50 mg placebo tablet, one 100 mg E5555 tablet, and one 100 mg placebo tablet, once daily for 12 weeks.
  Interventions: Drug: E5555; Drug: Placebo
- 3 (Active Comparator): Participants will receive one 50 mg placebo tablet and two 100 mg E5555 tablets, once daily for 12 weeks.
  Interventions: Drug: E5555; Drug: Placebo
- 4 (Placebo Comparator): Participants will receive one 50 mg placebo tablet and two 100 mg placebo tablets, once daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: E5555
  Arms: 1; 2; 3
Drug: Placebo

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled study to determine the safety and tolerability of E5555 in subjects with Acute coronary syndrome (ACS).

ELIGIBILITY:
INCLUSION CRITERIA:

1. Males or Females, 45 - 80 years of age
2. Presenting with features of non-ST segment elevation ACS (unstable angina or Myocardial infarction without persistent ST elevation). and at least one of the following two criteria on admission: Cardiac enzymes≥ ULN for the local institution OR ECG changes compatible with ischemia
3. Randomisation possible within 24 hours of the onset of the most recent symptomatic episode.

EXCLUSION CRITERIA:

1. History of acquired or congenital bleeding disorder, coagulopathy or platelet disorder, or history of pathological bleeding within the last 6 months
2. History of intracranial bleeding, history of hemorrhagic retinopathy, history of recent ischemic stroke or transient ischemic attack, or known structural cerebral vascular lesion
3. Recent trauma, major surgery, Percutaneous coronary intervention or coronary artery surgery
4. Clinically significant haematological, hepatic or renal abnormalities
5. Patients with some specific ST-segment changes, severe congestive heart failure or uncontrolled cardiac arrhythmias at baseline
6. Recent significant (as determined by the investigator) cardiovascular events

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2007-10; Primary Completion 2009-04 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | Up to 16 weeks

SECONDARY OUTCOMES:
Incidence of Major Adverse Cardiovascular Events; Platelet Aggregation Inhibition; Holter Monitoring. Exploratory Outcome Measure: effects on endovascular inflammatory processes | Up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rafal Ziecina, MD, Study Director — Eisai Limited
Locations (2):
- Beloit Clinic, SC, Beloit, Wisconsin, United States
- Royal Brompton Hospital, London, United Kingdom

REFERENCES:
- [Derived] O'Donoghue ML, Bhatt DL, Wiviott SD, Goodman SG, Fitzgerald DJ, Angiolillo DJ, Goto S, Montalescot G, Zeymer U, Aylward PE, Guetta V, Dudek D, Ziecina R, Contant CF, Flather MD; LANCELOT-ACS Investigators. Safety and tolerability of atopaxar in the treatment of patients with acute coronary syndromes: the lessons from antagonizing the cellular effects of Thrombin-Acute Coronary Syndromes Trial. Circulation. 2011 May 3;123(17):1843-53. doi: 10.1161/CIRCULATIONAHA.110.000786. Epub 2011 Apr 18. PMID 21502577